CLINICAL TRIAL: NCT02372682
Title: Shear Wave Sonoelastography for the Noninvasive Evaluation of Hepatic Fibrosis in the Pediatric Population
Brief Title: Shear Wave Sonoelastography in Pediatric Liver Fibrosis
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Shannon G. Farmakis, M.D., Assistant Professor, St. Louis University
Other Study IDs: 25138
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Sonoelastography; Elastography; Elastograms; Liver Fibrosis; Hepatic Fibrosis; Cirrhosis; Pediatrics
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Test: Any pediatric patient (0-18 years of age) with known liver disease in whom a liver biopsy is to be performed as standard of care to assess the degree of fibrosis will also undergo an abdominal ultrasound to evaluate the liver.
  Underlying diagnoses include but are not limited to biliary atresia, congenital fibrosis-cholestasis, Alagille syndrome, Caroli's disease, choledochal cyst, alpha-1-antitrypsin deficiency, progressive familial intrahepatic cholestasis (PFIC), viral hepatitis, glycogenosis, fructosemia, Wilson disease, cystic fibrosis, autosomal recessive polycystic kidney disease (ARPCKD), mesenterico-caval shunt, post liver transplant, and nonalcoholic steatohepatitis (NASH).
  Interventions: Device: Shear wave sonoelastography
- Control: Any pediatric patient (0-18 years of age) undergoing evaluation with an abdominal ultrasound as standard of care for evaluation for a diagnosis other than liver disease and in whom the US shows a normal liver, gallbladder, pancreas, spleen, and biliary tree will then be asked to enroll in the research study by undergoing shear wave elastography.
  Interventions: Device: Shear wave sonoelastography

INTERVENTIONS:
Device: Shear wave sonoelastography — Sonoelastography is to be performed on the liver.

SUMMARY:
Reliable methods of evaluating liver fibrosis using noninvasive techniques in the pediatric population are limited and inconclusive. Liver biopsy remains the gold standard; however, it requires sedation in pediatric patients, has a risk of hemorrhage, and provides unreliable results secondary to sampling error. Sonoelastography is a new method of evaluating liver disease that eliminates these pitfalls. There are 3 types of quantitative sonoelastography currently in use.

Transient elastography is a non-imaging based technique used in adults to measure liver fibrosis in which a mechanical vibrator creates a low-frequency wave causing shear stress in the liver at a fixed depth. This technique does not work in small livers and, therefore, is not appropriate for pediatric patients.

Acoustic Radiation Force Impulse Imaging (ARFI) and Shear Wave Imaging (SWE) use real-time ultrasonography and administer focused high-intensity, short-duration pulses to produce shear waves in the liver tissue. ARFI calculates the degree of tissue displacement and creates an elastogram or measurement of the stiffness of the sampled liver tissue without corresponding images. It is limited since only a small sample or region of interest (ROI) can be obtained, and it is unable to provide a corresponding elasticity map of the tissue.

SWE is the newest elastography technique. It measures tiny displacements of tissue in a larger ROI with corresponding ultrasound images which provides a side by side image of the liver and color-coded elasticity map of the sampled tissue. Advantages include a larger ROI and simultaneous viewing of the selected region of interest which provides better anatomic detail with a corresponding color map of the tissue elasticity which may result in more accurate scoring of the stage of fibrosis.

There are a few studies of ARFI in the pediatric population. Studies using SWE for evaluation of liver fibrosis are also few, and, all but one in adults. However, these studies have shown it to be an accurate method for liver fibrosis staging. Use of SWE in assessing liver fibrosis in pediatric patients may represent an accurate noninvasive alternative to liver biopsy in evaluating liver fibrosis as well as avoid the use of sedation.

DETAILED DESCRIPTION:
The evaluation of pediatric liver disease continues to be a major focus of research both in well-characterized liver diseases and in liver fibrosis secondary to obesity. The degree of fibrosis is generally well-accepted as both a measurement of disease severity and a prognostic indicator. Unfortunately, the current gold standard to assess fibrosis remains a liver biopsy, which, in addition to anesthesia risks and sampling errors, can result in profound hemorrhage, infections, and even mortality. Standard and reliable noninvasive biomarkers of hepatic fibrosis in the pediatric population are greatly needed. Sonoelastography has emerged as a method of evaluating liver disease. Three methods of quantitative sonoelastography are currently in use.

Transient elastography is an M-mode based sonographic technique in which a mechanical vibrator creates a low-frequency wave causing shear stress in the tissue at a fixed depth in the target tissue. It has gained widespread use in evaluation of liver fibrosis in the adult population (Fibroscan); however, its use has great limitations in the pediatric population as it does not use real-time ultrasonography (B mode) and has a fixed depth in which the measurement is taken. The lack of real-time imaging makes it impossible to accurately select an area for appropriate sampling, and the fixed depth is not appropriate for very young children with smaller livers. Also, the shock wave that is administered has not been tailored for use in young children. Furthermore, this technique is very unreliable in patients that are obese or who have ascites.

Other methods of sonoelastography include Acoustic Radiation Force Impulse Imaging (ARFI) and Shear Wave Elastography (SWE). The latter is also known as supersonic shear wave imaging. Both of these techniques use real-time ultrasonography and administer focused high-intensity, short-duration (acoustic radiation) pulses to produce shear waves in the target tissue. Neither technique is limited by the presence of ascites as the shear waves propagate through the fluid. ARFI uses a single pushing beam to generate the shear waves, and the propagation of those shear waves are monitored using conventional pulse-echo ultrasound at various off-axis lateral locations. The speed of the shear wave in the tissue is determined by collecting the displacement through time. This principle of elastography is based on the Young modulus using the formula: E=3ρѴ2 (E elasticity's modulus, Ѵ speed, ρ density of the tissue). The degree of tissue displacement is then used to create an elastogram. Limitations of ARFI include a small selected region of interest (ROI) (10 mm x 5 mm), it is a 1-dimensional technique, and it is unable to provide a corresponding elasticity map of the tissue. The latter also prevents retrospective evaluations of the tissue elasticity.

SWE is the newest elastography technique. It works by generating a localized radiation force that travels faster down the acoustic axis than the shear wave speed producing tiny, almost simultaneous, displacements in the tissues at all positions along the acoustic axis. The generated shear wave is shaped like a cone or fan, known as the Mach cone. An ultrafast sonography is then performed which provides a side-by-side greyscale image and color-coded elasticity map of the tissue in the ROI. The ROI is displayed in real time B-mode imaging and, thus, represents a 2-dimensional technique. Advantages include a larger, fan-shaped ROI (up to 50mm x 50mm), and the acquisition of a quantitative map of liver tissue stiffness with corresponding greyscale ultrasound image. As a result, simultaneous viewing of the selected region of interest provides better anatomic detail with a corresponding color map of the tissue elasticity which may result in more accurate scoring of the stage of fibrosis. The presence of a color map also allows for retrospective analysis.

Only a few studies have begun to use ARFI to analyze liver fibrosis in the pediatric population. Studies using SWE for evaluation of liver fibrosis are also limited and all but one have been performed in adults; however, early studies have shown it to be an accurate method for liver fibrosis staging. Tutar, et al safely performed a study using SWE in pediatric patients in Turkey. No dedicated pediatric studies have been performed in the United States, as the technology was just recently approved for use in adults by the FDA. The use of this device in pediatrics represents an off-label use. That being said, SWE has safety considerations that are similar to Doppler mode which is a standard ultrasound technology performed in pediatric patients of all ages. While it has a higher thermal index than routine B-mode ultrasound, it is measured to be within the safety limits set by the American Institute of Ultrasound in Medicine (AIUM).

ELIGIBILITY:
Inclusion Criteria:

* Any pediatric patient (0-18 years of age) with known liver disease with plans to undergo a liver biopsy within 1 month of ultrasound exam. Underlying diagnoses include biliary atresia, congenital fibrosis-cholestasis, Alagille syndrome, Caroli's disease, choledochal cyst, alpha-1-antitrypsin deficiency, progressive familial intrahepatic cholestasis (PFIC), viral hepatitis, glycogenosis, fructosemia, Wilson disease, cystic fibrosis, autosomal recessive polycystic kidney disease (ARPCKD), mesenterico-caval shunt, post liver transplant, and nonalcoholic steatohepatitis (NASH). Written informed consent from parent or legal guardian. Written informed assent from the child.

Exclusion Criteria:

* Inconclusive biopsy results. Patient not cooperative for the ultrasound exam. Failure to give informed consent. No biopsy results within allotted time frame. Poor acoustic window in which to perform sonoelastography.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The test population is pediatric patient (0-18 years of age) with known liver disease with plans to undergo a liver biopsy within 1 month of ultrasound exam. Underlying diagnoses include but are not limited to biliary atresia, congenital fibrosis-cholestasis, Alagille syndrome, Caroli's disease, choledochal cyst, alpha-1-antitrypsin deficiency, progressive familial intrahepatic cholestasis (PFIC), viral hepatitis, glycogenosis, fructosemia, Wilson disease, cystic fibrosis, autosomal recessive polycystic kidney disease (ARPCKD), mesenterico-caval shunt, post liver transplant, and nonalcoholic steatohepatitis (NASH).
  The control population is any pediatric patient (0-18 years of age) undergoing an abdominal ultrasound for reasons other than liver disease and in whom the US shows a normal liver, gallbladder, pancreas, spleen, and biliary tree.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Farmakis, MD, Principal Investigator — Assistant Professor, Saint. Louis University
Locations (1):
- St. Louis University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test: Any pediatric patient (0-18 years of age) with known liver disease in whom a liver biopsy is to be performed as standard of care to assess the degree of fibrosis will also undergo an abdominal ultrasound to evaluate the liver.
  Underlying diagnoses include but are not limited to biliary atresia, congenital fibrosis-cholestasis, Alagille syndrome, Caroli's disease, choledochal cyst, alpha-1-antitrypsin deficiency, progressive familial intrahepatic cholestasis (PFIC), viral hepatitis, glycogenosis, fructosemia, Wilson disease, cystic fibrosis, autosomal recessive polycystic kidney disease (ARPCKD), mesenterico-caval shunt, post liver transplant, and nonalcoholic steatohepatitis (NASH).
  Shear wave sonoelastography: Sonoelastography is to be performed on the liver.
Period: Overall Study
Arm/Group | Test | Control
Started | 78 | 93
Completed | 70 | 79
Not Completed | 8 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Control | Total
Number analyzed (Participants) | 70 | 79 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (6.0) | 11.0 (4.5) | 10.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 55 | 89
  Male | 36 | 24 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.5 (8.4) | 19.7 (4.8) | 23.5 (13.1)

OUTCOME MEASURES:

1. Primary Outcome: 2D-SWE Measurements' Capability of Predicting Stages of Fibrosis Based on METAVIR Scoring System
Description: METAVIR score is a tool used to measure fibrosis as seen on liver biopsy and scored to describe liver disease progress and prognosis.
Time Frame: 2 years
Measure: Number; unit: percentage of exams
Groups:
- Controls+METAVIR 0: Controls+METAVIR 0 (no portal fibrosis)
- METAVIR F1: portal fibrosis without septa
- METAVIR F2: portal fibrosis with few septa
- METAVIR F3: septal fibrosis without cirrhosis
Arm/Group | Controls+METAVIR 0 | METAVIR F1 | METAVIR F2 | METAVIR F3
Number analyzed (Participants) | 112 | 16 | 11 | 10
percentage of exams
  Sensitivity | NA — For pts without liver disease/fibrosis to be detected, no correlation can be made to determine sensitivity | 96.9 | 95.2 | 1.00
  Specificity | NA — For pts without liver disease/fibrosis to be detected, no correlation can be made to determine specificity | 80.2 | 70.7 | 64.1
  PPV | NA — For pts without liver disease/fibrosis to be detected, no correlation can be made to determine PPV | 66.0 | 42.6 | 21.3
  NPV | NA — For pts without liver disease/fibrosis to be detected, no correlation can be made to determine NPV | 98.5 | 98.5 | 1.00

2. Primary Outcome: 2D-SWE Measurements' Capability of Predicting Stages of Fibrosis Based on Ishak Scoring System
Description: Ishak is a tool used to evaluate liver fibrosis via liver biopsy to report severity and prognosis of liver disease, specifically hepatitis.
Time Frame: 2 years
Measure: Number; unit: percentage of exams
Groups:
- Control + Ishak 0: Control + Ishak 0 (no fibrosis)
- Ishak 1: Fibrous expansion of some portal areas, with or without short fibrous septa
- Ishak 2: Fibrous expansion of most portal areas, with or without short fibrous septa
- Ishak 3: Fibrous expansion of most portal areas, with occasional portal to portal (P-P) bridging
- Ishak 4: Fibrous expansion of portal areas, with marked bridging (portal to portal (P-P) as well as portal to central (P-C)
Arm/Group | Control + Ishak 0 | Ishak 1 | Ishak 2 | Ishak 3 | Ishak 4
Number analyzed (Participants) | 111 | 14 | 3 | 14 | 7
percentage of exams
  Sensitivity | NA — For pts without liver disease/fibrosis to be detected, no correlation can be made to determine sensitivity | 93.8 | 95.8 | 95.2 | 100.0
  Specificity | NA — For pts without liver disease/fibrosis to be detected, no correlation can be made to determine specificity | 79.0 | 73.0 | 70.7 | 62.3
  PPV | NA — For pts without liver disease/fibrosis to be detected, no correlation can be made to determine PPV | 63.8 | 48.9 | 42.6 | 14.9
  NPV | NA — For pts without liver disease/fibrosis to be detected, no correlation can be made to determine NPV | 96.9 | 98.5 | 98.5 | 100.0

ADVERSE EVENTS:
Time Frame: 30 minutes.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/79
Other Adverse Events (participants affected / at risk) | 0/70 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GE - Contract states: "The Institution [SLU/PI] is free to publish or present the results of the Study. The Institution agrees to provide Company with a copy of the published manuscript. Company's support will be acknowledged in all such publications or presentations." Thrasher - No restrictions on publication Society of Pediatric Radiology - Manuscripts must be first submitted to SPR annual Meeting and/or to Pediatric Radiology journal, to be considered for publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT02372682/Prot_SAP_000.pdf